CLINICAL TRIAL: NCT01920867
Title: Bone Marrow Derived Stem Cell Ophthalmology Treatment Study
Brief Title: Stem Cell Ophthalmology Treatment Study
Acronym: SCOTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: MD Stem Cells (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICMS-2013-0019.
Record Dates: First submitted 2013-08-08; First posted 2013-08-12 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Retinal Disease; Macular Degeneration; Hereditary Retinal Dystrophy; Optic Nerve Disease; Glaucoma
Keywords: Stem Cells; Bone Marrow Derived Stem Cells; BMSC; BMC (Bone Marrow Cell); Mesenchymal Stem Cells; MSC; Eye Disease; Eye Stem Cells; Ophthalmology; Ophthalmic Disease; Retina; Retinal Disease; Macular Degeneration; Age Related Macular Degeneration; Myopic Macular Degeneration; Geographic Atrophy; Dry Macular Degeneration; Wet Macular Degeneration; Retinal Atrophy; Retinal Dystrophy; Hereditary Retinal Dystrophy; Retinitis Pigmentosa; Stargardt Disease; Cone Dystrophy; Cone Rod Dystrophy; Maculopathy; Optic Nerve Disease; Optic Nerve Atrophy; Optic Atrophy; Ischemic Optic Neuropathy; Optic Nerve Damage; Optic Nerve Compression; Compressive Optic Neuropathy; Devics Syndrome
MeSH Terms: conditions — Retinal Diseases; Macular Degeneration; Optic Nerve Diseases; Glaucoma; Eye Diseases; Geographic Atrophy; Wet Macular Degeneration; Retinal Dystrophies; Retinitis Pigmentosa; Stargardt Disease; Cone Dystrophy; Cone-Rod Dystrophies; Optic Atrophy; Optic Neuropathy, Ischemic; Optic Nerve Injuries; Neuromyelitis Optica | interventions — Immunoglobulins, Intravenous; Jupiter; Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- RB, ST, IV (Active Comparator): Injections of BMSC retrobulbar (RB), subtenon (ST) and intravenous (IV)
  Interventions: Procedure: RB (Retrobulbar); Procedure: ST (Subtenon); Procedure: IV (Intravenous)
- RB, ST, IV, IVIT (Active Comparator): Injections of BMSC retrobulbar, subtenon, intravenous and intravitreal ( IVIT )
  Interventions: Procedure: RB (Retrobulbar); Procedure: ST (Subtenon); Procedure: IV (Intravenous); Procedure: IVIT (Intravitreal)
- RB, ST, IV, IO (Active Comparator): Injection of BMSC retrobulbar, subtenon, intravenous and intraocular (IO) with vitrectomy
  Interventions: Procedure: RB (Retrobulbar); Procedure: ST (Subtenon); Procedure: IV (Intravenous); Procedure: IO (Intraocular)

INTERVENTIONS:
Procedure: RB (Retrobulbar) — Retrobulbar injection of Bone Marrow Derived Stem Cells (BMSC)
  Other Names: Retrobulbar injection of stem cells
Procedure: ST (Subtenon) — Subtenon injection of Bone Marrow Derived Stem Cells (BMSC)
  Other Names: Subtenon injection of stem cells
Procedure: IV (Intravenous) — Intravenous injection of Bone Marrow Derived Stem Cells (BMSC)
  Other Names: Intravenous injection of stem cells
Procedure: IVIT (Intravitreal) — Intravitreal injection of Bone Marrow Derived Stem Cells (BMSC)
  Other Names: Intravitreal injection of stem cells
  Arms: RB, ST, IV, IVIT
Procedure: IO (Intraocular) — Intraocular injection of Bone Marrow Derived Stem Cells (BMSC) with vitrectomy prior to intraocular injection. For example, may include larger amount of stem cells in the intravitreal cavity, intraneuronal injections or subretinal injections of stem cells.
  Other Names: Intraocular injection of stem cells with vitrectomy
  Arms: RB, ST, IV, IO

SUMMARY:
This study will evaluate the use of autologous bone marrow derived stem cells (BMSC) for the treatment of retinal and optic nerve damage or disease. http://mdstemcells.com/scots-ii/

DETAILED DESCRIPTION:
Eyes with loss of vision from retinal or optic nerve conditions generally considered irreversible will be treated with a combination of injections of autologous bone marrow derived stem cells isolated from the bone marrow using standard medical and surgical practices. Retinal conditions may include degenerative, ischemic or physical damage ( examples may include macular degeneration, hereditary retinal dystrophies such as retinitis pigmentosa, stargardt, non-perfusion retinopathies, post retinal detachment. Optic Nerve conditions may include degenerative, ischemic or physical damage ( examples may include optic nerve damage from glaucoma, compression, ischemic optic neuropathy, optic atrophy ). Injections may include retrobulbar, subtenon, intravitreal, intraocular, subretinal and intravenous. Patients will be followed for 12 months with serial comprehensive eye examinations including relevant imaging and diagnostic ophthalmic testing.

ELIGIBILITY:
Inclusion Criteria:

* Have objective, documented damage to the retina or optic nerve unlikely to improve OR
* Have objective, documented damage to the retina or optic nerve that is progressive
* AND have less than or equal to 20/40 best corrected central visual acuity in one or both eyes AND/OR an abnormal visual field in one or both eyes.
* Be at least 3 months post-surgical treatment intended to treat any ophthalmologic disease and stable.
* If under current medical therapy ( pharmacologic treatment) for a retinal or optic nerve disease be considered stable on that treatment and unlikely to have visual function improvement ( for example, glaucoma with intraocular pressure stable on topical medications but visual field damage ).
* Have the potential for improvement with BMSC treatment and be at minimal risk of any potential harm from the procedure.
* Be over the age of 18
* Be medically stable and able to be medically cleared by their primary care physician or a licensed primary care practitioner for the procedure. Medical clearance means that in the estimation of the primary care practitioner, the patient can reasonably be expected to undergo the procedure without significant medical risk to health.

Exclusion Criteria:

* Patients who are not capable of an adequate ophthalmologic examination or evaluation to document the pathology.
* Patients who are not capable or not willing to undergo follow up eye exams with the principle investigator or their ophthalmologist or optometrist as outlined in the protocol.
* Patients who are not capable of providing informed consent.
* Patients who may be at significant risk to general health or to the eyes and visual function should they undergo the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 1 day to 12 months
  Best corrected visual acuity will be measured with Snellen Eye Chart and the ETDRS (Early Treatment Diabetic Retinopathy Study)Eye Chart when available at each post- procedure visit. Intervals at minimum will be first post- procedure day,then 3 months, 6 months and 12 months post-procedure day. Recommended visit 1 month post -procedure day.

SECONDARY OUTCOMES:
Visual fields | 1 day to 12 months
  Visual fields will be evaluated with automated perimetry during post- procedure visits as needed and specifically at 6 months and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Levy, MD, Study Director — MD Stem Cells; Jeffrey Weiss, MD, Principal Investigator — MD Stem Cells
Locations (1):
- MD Stem Cells, Westport, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weiss JN, Levy S, Malkin A. Stem Cell Ophthalmology Treatment Study (SCOTS) for retinal and optic nerve diseases: a preliminary report. Neural Regen Res. 2015 Jun;10(6):982-8. doi: 10.4103/1673-5374.158365. PMID 26199618
- [Result] Weiss JN, Levy S, Benes SC. Stem Cell Ophthalmology Treatment Study (SCOTS) for retinal and optic nerve diseases: a case report of improvement in relapsing auto-immune optic neuropathy. Neural Regen Res. 2015 Sep;10(9):1507-15. doi: 10.4103/1673-5374.165525. PMID 26604914
- [Result] Weiss JN, Benes SC, Levy S. Stem Cell Ophthalmology Treatment Study (SCOTS): improvement in serpiginous choroidopathy following autologous bone marrow derived stem cell treatment. Neural Regen Res. 2016 Sep;11(9):1512-1516. doi: 10.4103/1673-5374.191229. PMID 27857759
- [Derived] Kasetty MA, Hedges TR 3rd, Witkin AJ. BILATERAL EPIRETINAL MEMBRANE FORMATION AFTER INTRAVITREAL INJECTIONS OF AUTOLOGOUS MESENCHYMAL STEM CELLS. Retin Cases Brief Rep. 2022 Sep 1;16(5):561-564. doi: 10.1097/ICB.0000000000001032. PMID 32568958
- [Derived] Weiss JN, Levy S, Benes SC. Stem Cell Ophthalmology Treatment Study (SCOTS): bone marrow-derived stem cells in the treatment of Leber's hereditary optic neuropathy. Neural Regen Res. 2016 Oct;11(10):1685-1694. doi: 10.4103/1673-5374.193251. PMID 27904503
- See also: The Role of Patient Funded Clinical Research in Advancing Medical Care — https://mdstemcells.com